CLINICAL TRIAL: NCT03518788
Title: Randomized Clinical Trial to Evaluate the Efficacy of the Permanent Thoracic Catheter (Pleur-X) Towards Pleurodesis in Thoracoscopy in the Treatment of Malignant Pleural Effusion
Brief Title: Malignant Pleural Effusion: Pleur-X vs. Chemical Pleurodesis in VATS
Acronym: Pleur-X
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rolf Inderbitzi (Other)
Collaborators: Clinical Trial Unit Ente Ospedaliero Cantonale (Other)
Responsible Party: Sponsor-Investigator, Rolf Inderbitzi, Head of thoracic surgery department, Ente Ospedaliero Cantonale, Bellinzona
Organization: Ente Ospedaliero Cantonale, Bellinzona (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ORBV-CHIR-001
Record Dates: First submitted 2018-04-06; First posted 2018-05-08 (Actual); Last update posted 2018-05-08 (Actual); Status verified 2018-04

CONDITIONS: Malignant Pleural Effusion
MeSH Terms: conditions — Pleural Effusion, Malignant | interventions — Pleurodesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pleur-X (Experimental): Placement of a permanent drainage under local anesthesia
  Interventions: Procedure: Pleur-X
- pleurodesis (Experimental): Pleurodesis with talc in VATS
  Interventions: Procedure: Pleurodesis

INTERVENTIONS:
Procedure: Pleur-X — Permanent drainage
  Arms: Pleur-X
Procedure: Pleurodesis — Pleurodesis with talc in permanent VATS
  Arms: pleurodesis

SUMMARY:
This is a prospective randomized study whose aim is to compare the efficacy of the permanent thoracic catheter (Pleur-X) versus chemical pleurodesis in videothoracoscopy (VATS) in the treatment of malignant pleural effusion at the first diagnosis.Patients with malignant pleural effusion for whom there is indication of surgery and who agree to participate in the study will be randomized 1: 1 in the Pleur-X arm (arm 1) or in the chemical pleurodesis arm (arm 2).

The arm 1 provides for the installation of a permanent drainage under local anesthesia while the arm 2 provides a pleurodesis with talc in VATS under general anesthesia.

Both procedures are standard of care.

DETAILED DESCRIPTION:
Before the study procedure the patients will be requested to perform some examination as physical and radiological examination. Patients will also complete questionnaires for quality of life assessment (EORTC QLQ 30) and symptoms (VAS for pain). Patients will then be randomized into one of the two arms.

For patients included in arm 1, a permanent drainage (Pleur-X) is provided under local anesthesia performed on an outpatient basis while for patients included in arm 2 a pleurodesis with talc in VATS is planned under general anesthesia. Arm 2 patients will be hospitalized for 5 days.

Patients will then be followed up to 3 months after surgery. During this period a medical examination will be required at 1 week, 4 weeks and 3 months after the intervention during which the patient will be asked to complete questionnaires for the evaluation of quality of life (EORTC QLQ 30) and symptoms (VAS for pain ). A chest radiograph will be performed after four weeks to evaluate the primary parameter. Adverse events will be collected throughout the study period.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years, <80 years
* First diagnosis of malignant pleural effusion
* Indication to treat the malignant pleural effusion with surgery
* Informed informed consent

Exclusion Criteria:

* Previous surgeries on the same hemitorace
* Pregnant women
* Trapped lung syndrome
* Patients with estimated life expectancy < 4-8 weeks

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Estimated)
Dates: Start 2018-01-25 (Actual); Primary Completion 2020-03-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Success rate of the treatment with VPM | 4 weeks
  Evaluate the success rate of the treatment with VPM with radiological examination

SECONDARY OUTCOMES:
Adverse Event | 3 months
  Evaluate the tollerability of both procedures collecting adverse events
Quality of live | 3 months
  quality of live will be determined with the evaluation of the EORTC QLQ 30 questionnaire
Pain scale | 3 months
  Pain will be evaluated with the Visual Analogue Scale (VAS) where the score of 0 is no pain while the score 10 is very painfull

CONTACTS AND LOCATIONS:
Overall Officials: Rolf Inderbitzi, MD, Study Director — Ente Ospedaliero Cantonale, Bellinzona
Locations (1):
- Ospedale San Giovanni, Bellinzona, Switzerland